CLINICAL TRIAL: NCT06244784
Title: Effectiveness of an Interventional Intervention in Improving the Work Environment of Nurses and Nursing Assistants in the Hospital
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Estel Curado Santos, RN, MsN, PhDc, Universitat Internacional de Catalunya
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INF-2022-01; 20212013 (Registry Identifier: Hospital General de Granollers); 02-23-305-060 (Registry Identifier: Consocri Sanitari de Terrassa); PR-551/2022 (Other Grant/Funding Number: Official College of Nurses of Barcelona)
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Healthy Work Environment; Burnout; Intention to Leave; Engagement
Keywords: Healthy Work Environment; Burnout; Intent to leave; Engagement; Educational intervention; Nursing
MeSH Terms: conditions — Burnout, Psychological | interventions — Nurses; Nursing Assistants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive the training course on healthy work environment
  Interventions: Behavioral: effectiveness of a training course on a healthy work environment for nurses and nursing assistants in a hospital
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: effectiveness of a training course on a healthy work environment for nurses and nursing assistants in a hospital — Once the participants have been included in the study, they will be assigned to each group; control group and intervention group by convenience sampling. Baseline data will be collected in both groups. At this time, questionnaires will be collected in both populations and focus groups will be conducted in the professionals assigned to both groups. Once the data have been obtained, the intervention group will conduct the training course.
  After the training, data will be collected again at three different times: 1) Right after the training: questionnaires and focus group will be collected from intervention group professionals; 2) 6 months after the training: questionnaires will be collected from control group and intervention group; 3) 12 months after the training: questionnaires will be collected and focus groups will be conducted in both groups.
  Arms: Intervention Group

SUMMARY:
The goal of this interventional study is to evaluate the effectiveness of a training course on a healthy work environment for nurses and nursing assistants in a hospital. The main questions it aims to answer are:

* To evaluate the effectiveness of a training course on a healthy work environment
* To know the perception of nursing and nursing assistants on what is needed to have a healthy work environment, what elements it should contain and whether it has changed after the course has been completed

Participants in the intervention group will receive the training course and the control group will not. Researchers will compare intervention group with control group to see if the training course on healthy work environment is effective.

DETAILED DESCRIPTION:
Concurrent mixed study consisting of different phases in which the qualitative and quantitative parts will be interspersed. The qualitative part will include focus groups, and the quantitative part will be a controlled non-randomised experimental study by convenience sampling according to hospital unit and professional category (nurses and nursing assistants). Multicenter study carried out at Hospital General de Granollers and the Consorci Sanitari de Terrassa in nursing professionals and nursing assistants with one year of experience working in the hospital in any of the hospitalization services or special services. Once the subjects have been included in the study, they will be assigned in each group (control group and intervention group) through a stratification by quotas following the same criteria as in the sampling. The intervention group will receive training (n=56), and the control group will not (n=112). The training will be based on the American Association of Critical Care Nurses standards on a healthy work environment. In both groups, the same data will be collected at different times (before and just after the training, at 6 months and 12 months post-training). The focus groups will not be conducted in the control group after the training. Work environment, burnout, intention to leave the job and staff engagement will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary acceptance to participate in the study
* Having worked at least one year in the hospital

Exclusion Criteria:

* Nursing supervisors/nursing assistants or people with management positions
* Professionals working in more than one care center
* Professionals working in the outpatient area

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Work Environment (1) | 1year
  The Practice Environment Scale-Nursing Work Index (PES-NWI) will be used to assess the work environment. The PES-NWI is used to measure day-to-day aspects of organizational culture and climate, and is more frequently used in European studies. The PES-NWI is Likert-type with scores from 1 to 4 (strongly disagree - strongly agree). Three category variable indicating favorable, mixed, or unfavorable practice environments: favorable = four or more subscale means exceed 2.5; mixed = two or three subscale means exceed 2.5; unfavorable = zero or one subscales exceed 2.5.
Work Environment (2) | 1year
  The American Association of Critical Care Nurses (AACN) questionnaire will be used to assess the work environment. The AACN questionnaire is much broader and covers other aspects related to the work environment. The AACN scoring guidelines for the assessment are: 1.00-2.99 - Needs Improvement 3.00-3.99 - Good 4.00-5.00 - Excellent.

SECONDARY OUTCOMES:
Burnout | 1 year
  Questionnaire for the Assessment of Job Burnout Syndrome (CESQT) will be used to evaluate the burnout syndrome in professionals who care for people.
Engagement | 1 year
  Utrecht work engagement scale (UWES) will be use to assess the engagement. The UWES contais 17 items; 6 items in reference to vigor (item 1, ,4, 8, 12, 15, 17), 5 items to dedication (item 2, 5, 7, 7, 10 13) and 6 items to absorption (item 3, 6, 9, 11, 14, 16). It is a frequency scale with 6 response options from 0 (never) to every day (6).
Intention to leave | 1 year
  The American Association of Critical Care Nurses questionnaire will be used to assess the intention to leave of participants.
Focus groups | 1 year
  Professionals participating in the study will be invited to collaborate in focus groups depending on the time of the study. These will take place at different times and will have different objectives. Before the intervention (control group and intervention group), they will focus on what they consider to be a healthy work environment and what elements they identify it should contain. After the intervention (only intervention group), we will explore how their perception of what a healthy work environment is has changed. At 12 months (control group and intervention group), we will explore whether there has been any change during this time in the work environment and the perceptions about the actions they consider that the institution and/or professionals could take to improve the work environment.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital General de Granollers, Granollers, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona

IPD SHARING:
Plan to Share IPD: No